CLINICAL TRIAL: NCT04688294
Title: The Bio-Clinical Effects of the (Sacubitril-Valsartan) Combination on Patients With Chronic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amir Safwat (Other)
Responsible Party: Sponsor-Investigator, Amir Safwat, Teaching assistant, Suez Canal University
Organization: Suez Canal University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/2019
Record Dates: First submitted 2020-12-19; First posted 2020-12-29 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril/valsartan (Experimental): Group 30 patients will undergo treatment with sacubitril/valsartan combination according to guideline-directed medical therapy.
  Interventions: Drug: Sacubitril-Valsartan
- Valsartan (Active Comparator): Group 30 patients will undergo treatment with valsartan according to guideline-directed medical therapy.
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Sacubitril-Valsartan — 30 patients initially received Sacubitril/Valsartan at 24/26 mg twice daily orally then dose was doubled as tolerated every 2-4 weeks to reach the target maintenance dose 97 mg/103 mg twice daily
  Arms: Sacubitril/valsartan
Drug: Valsartan — 30 patients received valsartan, starting at a dose of 40 mg/day orally. The dose was then doubled every 1-2 weeks on the basis of their blood pressure to reach a dose of 160 mg once daily according to guideline-directed medical therapy.
  Arms: Valsartan

SUMMARY:
The aim of this study is to evaluate the bio-clinical effects of sacubitril/valsartan combination in treatment of patients with Congestive heart failure. Moreover, the investigators aim to evaluate side effects of this combination.

- The following parameters were determined at baseline and at end of the study at 6 months of the beginning.

1. New York Heart Association (NYHA) Class.
2. Frequency of hospitalization by acute exacerbation of CHF
3. NT-ProBNP
4. Left ventricular systolic function by Echocardiography

Moreover, the side effects of the drugs used during study was assessed by

1. Renal function (Serum creatinine) was performed every month till the end of the study.
2. Serum electrolytes (Potassium and Sodium) was performed every month till the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 - 60 years
2. Patients with chronic congestive heart failure class ( II-IV) symptoms according to New York Heart Association (NYHA) classification
3. Left Ventricular Ejection Fraction of 40% or less.
4. NT-proBNP level of at least ≥400 pg per milliliter
5. ACE-inhibitor or ARB therapy with stable dose for prior 4 weeks, equivalent to enalapril ≥ 10 mg/day.

Exclusion Criteria:

1. Patients with symptomatic hypotension.
2. Pregnant and nursing women
3. Systolic blood pressure < 100 mmHg at screening or < 95 mmHg at randomization
4. Patients with glomerular filtration rate <30 mL/min/1.73 m2
5. Patients with history of angioedema
6. Patients with unacceptable side effects with ACE-inhibitors or ARBs.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
change in NTproBNP plasma concentration | at baseline
  NTproBNP is a Biomarker used to assess severity of congestive heart failure)
change in NTproBNP plasma concentration | at 6 months
  NTproBNP is a Biomarker used to assess severity of congestive heart failure)
severity of congestive heart failure. | at baseline
  Ejection fraction
severity of congestive heart failure. | at 6 months
  Ejection fraction

SECONDARY OUTCOMES:
change in plasma potassium concentration | every month, up to 6 months
  plasma potassium (intracellular cation) concentration used to evaluate Sacubitril-Valsartan
change in serum sodium concentration | every month, up to 6 months
  serum sodium (extracellular cation) concentration used to evaluate Sacubitril-Valsartan
change in serum creatinine | every month, up to 6 months
  serum creatinine which is a byproduct of muscle protein metabolism is used to evaluate Sacubitril-Valsartan

CONTACTS AND LOCATIONS:
Locations (1):
- Wadi El-Neel Hospital, Cairo, Egypt